CLINICAL TRIAL: NCT06759142
Title: Analysis of Patients With Autosomal Dominant Polycystic Kidney
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ADPKD-TO2020
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Autosomal Dominant Polycystic Kidney; ADPKD
Keywords: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the study is to establish a database of clinical data and genetic data of patients diagnosed with ADPKD, with particular focus on those who have undertaken a specific therapy (Tolvaptan or Octreotide), afferent to the Integrated Renal Genetic Diseases Outpatient Clinic of the U.O. Nephrology, Dialysis and Transplantation of the Sant'Orsola-Malpighi Polyclinic directed by Prof. La Manna. In-depth analysis and comparison on clinical, laboratory and instrumental outcomes will be performed within this population.

A thorough personal and family history will be obtained, and once informed consent is obtained, data will be entered and updated during subsequent outpatient monitoring.

Attention is paid to the clinical course of the disease in relation to genetic variants (genotype-phenotype correlation) and treatments performed by patients, in order to monitor the progression of the disease to end-stage renal failure (ESRD) and the impact that specific therapy has on various parameters identified as indicating such progression. In particular, monitoring of the reduction in renal function, as assessed by creatinine, eGFR, 24-hour proteinuria, and urinary osmolarity values, with attention to comparing developmental trends toward ESDR between patients not receiving therapy and patients on specific therapy, and monitoring of the numerical and/or volumetric increase in renal cysts, as assessed by imaging comparison of the TKV value at the time of diagnosis of polycystic kidney disease and at subsequent re-evaluation, with attention to the extent of progression following the initiation of specific therapy, will be performed.

DETAILED DESCRIPTION:
The main objective of the study is to establish a database of clinical data and genetic data of patients diagnosed with ADPKD, with particular focus on those who have undertaken a specific therapy (Tolvaptan or Octreotide), afferent to the Integrated Renal Genetic Diseases Outpatient Clinic of the U.O. Nephrology, Dialysis and Transplantation of the Sant'Orsola-Malpighi Polyclinic directed by Prof. La Manna. In-depth analysis and comparison on clinical, laboratory and instrumental outcomes will be performed within this population.

A thorough personal and family history will be obtained, and once informed consent is obtained, data will be entered and updated during subsequent outpatient monitoring.

Attention is paid to the clinical course of the disease in relation to genetic variants (genotype-phenotype correlation) and treatments performed by patients, in order to monitor the progression of the disease to end-stage renal failure (ESRD) and the impact that specific therapy has on various parameters identified as indicating such progression. In particular, monitoring of the reduction in renal function, as assessed by creatinine, eGFR, 24-hour proteinuria, and urinary osmolarity values, with attention to comparing developmental trends toward ESDR between patients not receiving therapy and patients on specific therapy, and monitoring of the numerical and/or volumetric increase in renal cysts, as assessed by imaging comparison of the TKV value at the time of diagnosis of polycystic kidney disease and at subsequent re-evaluation, with attention to the extent of progression following the initiation of specific therapy, will be performed.

The secondary objectives of the study are:

1. cardiovascular monitoring, understood as analysis of the pressor profile, valvular and cerebral pathologies: special attention will be paid to the diagnosis and course of hypertension and its therapeutic management, the presence of valvulopathy and its course, the presence of aneurysmal changes in the cerebral circulation and its course
2. the monitoring of urologic complications associated with polycystic disease, such as stones, urinary tract infections, and episodes of macrohematuria.
3. the monitoring of other conditions associated with polycystic disease, such as hepatic involvement, considering cystic involvement by imaging and laboratory indices of damage, and presence of reported and/or objective bulking syndrome (presence of abdominal wall hernias)
4. monitoring of side effects of specific therapy: increased uricemia with possible need for therapeutic adjustment, acute liver damage, quality and severity of symptoms related to water loss with regard to Tolvaptan, quality and severity of gastrointestinal symptoms with regard to Octreotide. In both subgroups of patients on specific treatment, the possible need for momentary or permanent discontinuation of therapy will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age-matched subjects with a diagnosis of ADPKD defined on the basis of the Unified Criteria of Pei. Diagnosis in subjects with a positive family history is based on age-differentiated ultrasound criteria. The presence of a "total of 3 or more cysts" in subjects aged 18-39 years and "2 or more cysts in each kidney" in at-risk subjects aged 40-59 years are sufficient to make the diagnosis of ADPKD.In the absence of family history, the presence of more than 10 cysts per kidney on ultrasound is typically considered diagnostic. Where the picture appears unclear, and particularly where the diagnosis has a major fallout (related to family planning, renal donation, initiation of specific drug treatment), genetic confirmation is strongly recommended.
* Obtaining Informed Written Consent.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a definite diagnosis of ADPKD referred to the Integrated Renal Genetic Disease Outpatient Clinic of theTU.O. Nephrology, Dialysis and Transplantation of Policlinico Sant'Orsola-Malpighi directed by Prof La Manna from 01/01/2017 to 01/06/2025.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
To establish a database of clinical data and genetic data of patients diagnosed with ADPKD | 5 years
  The main objective of the study is to establish a database of clinical data and genetic data of patients diagnosed with ADPKD, with particular focus on those who have undertaken a specific therapy (Tolvaptan or Octreotide), afferent to the Integrated Renal Genetic Diseases Outpatient Clinic of the U.O. Nephrology, Dialysis and Transplantation of the Sant'Orsola-Malpighi Polyclinic directed by Prof. La Manna. In-depth analysis and comparison on clinical, laboratory and instrumental outcomes will be performed within this population.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano La Manna, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No